CLINICAL TRIAL: NCT00472680
Title: Nutritional Regulation of Bone - Aim 2
Brief Title: The Effect of Severe Weight Loss and Protein Intake on Bone
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding didn't support further recruitment
Sponsor: Rutgers University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sue A. Shapses, Ph.D., RD, Professor, Rutgers University
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG0082; 5R01AG012161 (NIH)
Record Dates: First submitted 2007-05-10; First posted 2007-05-14 (Estimated); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Weight Loss
Keywords: bone mass; calcium absorption; bone quality; fracture risk
MeSH Terms: conditions — Weight Loss | interventions — Caloric Restriction; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): High Dietary Protein
  Interventions: Behavioral: Caloric restriction, high protein; Behavioral: Nutrition Education
- 2 (Active Comparator): Normal Dietary Protein
  Interventions: Behavioral: Caloric restriction; normal protein; Behavioral: Nutrition Education

INTERVENTIONS:
Behavioral: Caloric restriction, high protein — Weight loss with higher protein (35%) intake
  Arms: 1
Behavioral: Caloric restriction; normal protein — Weight loss with normal level of protein (18%) intake
  Arms: 2
Behavioral: Nutrition Education — Participants will have the opportunity to speak with the dietitian about their diet by phone, or on-site twice per month

SUMMARY:
The purpose of this study is to learn whether the amount of dietary protein can influence bone health during the weight loss after weight loss surgery.

DETAILED DESCRIPTION:
It is unclear whether the amount of protein in the diet during caloric restriction influences bone density. This information is important for determining optimal nutrient requirements during weight loss. This study will examine usual and higher dietary protein intake during severe weight loss following weight loss surgery on bone turnover, mass and quality in women, with the hypothesis that higher protein intake will reduce bone turnover and loss, and/or prevent the changes in bone quality associated with severe weight loss in women ages 18 to 70 years.

Participants will be randomly assigned to one of 2 groups: A) weight loss with recommended level of protein intake, or B) weight loss with higher protein intake. A dietitian will provide instructions for a reduced calorie, well balanced diet throughout the 12-month study using a nutrition-education behavior- modification program. Participants will have the opportunity to speak with the dietitian about their diet by phone, or on-site twice per month. In addition they will be asked to take a daily vitamin/mineral supplement and, depending on their usual food intake, they may be asked to take a calcium tablet to meet the recommended intake throughout the study period. Bone, mineral, protein and lipid markers, and hormones that influence bones will be measured. These measurements will provide information about body composition (fat, muscle mass, and bone mineral density).

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18 to 70 who are undergoing gastric bypass surgery
* Must live in the geographic vicinity of Rutgers University

Exclusion Criteria:

* Currently on any medication known to influence calcium or bone metabolism, including HRT, or with evidence of diseases known to influence calcium metabolism (i.e. metabolic bone disease, hyperparathyroidism, untreated thyroid disease, significant immune, hepatic, or renal disease, significant cardiac disease [i.e., heart attack or stroke in the past 6 months., abnormal EKG], active malignancy or cancer therapy within the past year)
* History of kidney stones
* Weight gain or weight loss (5% of body wt) within 3 months prior to recruitment
* Participation in other investigational studies during the 12-month study period
* Usually have a very high or low intake of calcium (more than 1500 or less than 500 mg per day)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-03; Primary Completion 2015-05 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Changes in Bone mineral density and quality | one year

SECONDARY OUTCOMES:
Changes in serum and urine bone markers, hormones, and proteins | one year

CONTACTS AND LOCATIONS:
Overall Officials: Sue A. Shapses, PhD, RD, Principal Investigator — Rutgers University, Nutritional Sciences
Locations (1):
- Rutgers University, New Brunswick, New Jersey, United States

REFERENCES:
- [Background] Shapses SA, Riedt CS. Bone, body weight, and weight reduction: what are the concerns? J Nutr. 2006 Jun;136(6):1453-6. doi: 10.1093/jn/136.6.1453. PMID 16702302
- [Background] Riedt CS, Cifuentes M, Stahl T, Chowdhury HA, Schlussel Y, Shapses SA. Overweight postmenopausal women lose bone with moderate weight reduction and 1 g/day calcium intake. J Bone Miner Res. 2005 Mar;20(3):455-63. doi: 10.1359/JBMR.041132. Epub 2004 Nov 29. PMID 15746990
- [Background] Goode LR, Brolin RE, Chowdhury HA, Shapses SA. Bone and gastric bypass surgery: effects of dietary calcium and vitamin D. Obes Res. 2004 Jan;12(1):40-7. doi: 10.1038/oby.2004.7. PMID 14742841
- [Background] Riedt CS, Brolin RE, Sherrell RM, Field MP, Shapses SA. True fractional calcium absorption is decreased after Roux-en-Y gastric bypass surgery. Obesity (Silver Spring). 2006 Nov;14(11):1940-8. doi: 10.1038/oby.2006.226. PMID 17135609
- [Background] Sukumar D, Ambia-Sobhan H, Zurfluh R, Schlussel Y, Stahl TJ, Gordon CL, Shapses SA. Areal and volumetric bone mineral density and geometry at two levels of protein intake during caloric restriction: a randomized, controlled trial. J Bone Miner Res. 2011 Jun;26(6):1339-48. doi: 10.1002/jbmr.318. PMID 21611972
- [Derived] Ogilvie AR, Schlussel Y, Sukumar D, Meng L, Shapses SA. Higher protein intake during caloric restriction improves diet quality and attenuates loss of lean body mass. Obesity (Silver Spring). 2022 Jul;30(7):1411-1419. doi: 10.1002/oby.23428. Epub 2022 May 11. PMID 35538903